CLINICAL TRIAL: NCT03010280
Title: A Controlled, Randomized, Open Clinical Trial to Compare the Effect of Preoperatory Treatment With Immunonutrition vs Hyperproteic Nutritional Supplements on Postoperative Inflammation Markers in Patients Going Through Bariatric Surgery
Brief Title: Effect of Immunonutrition on Inflamatory Markers After Bariatric Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Instituto de Investigación Sanitaria de la Fundación Jiménez Díaz (Other)
Collaborators: Hospital Universitario Rey Juan Carlos (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: INMUNOBAR-HURJC-15/01
Record Dates: First submitted 2017-01-03; First posted 2017-01-05 (Estimated); Last update posted 2018-02-14 (Actual); Status verified 2017-08

CONDITIONS: Postoperative Complications
MeSH Terms: conditions — Postoperative Complications | interventions — Immunonutrition Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Immunonutrition (Experimental): Patients receiving a preoperative balanced energy high-protein formula, enriched with Omega - 3 fatty acids (Immunonutrition formula)
  Interventions: Dietary Supplement: Immunonutrition
- Balanced high-protein formula (Active Comparator): Patients receiving a preoperative balanced energy high-protein formula, without including Omega - 3 fatty acids
  Interventions: Dietary Supplement: Balanced high-protein formula

INTERVENTIONS:
Dietary Supplement: Immunonutrition — Balanced high-protein formula enriched with Omega-3 fatty acids. 200 ml of formula every 8 hours during 10 days preoperatively
  Arms: Immunonutrition
Dietary Supplement: Balanced high-protein formula — Balanced high-protein formula, without Omega-3 fatty acids. 200 ml of formula every 8 hours during 10 days preoperatively
  Arms: Balanced high-protein formula

SUMMARY:
A prospective randomized clinical trial of all the patients undergoing Roux - en-Y gastric bypass will be performed. Patients will be randomly assigned into 2 groups: those patients receiving a preoperative balanced energy high-protein formula (group 1) and those receiving preoperative Immunonutrition (group 2). Changes between groups in acute inflamatory markers, pain, postoperative septic complications and lenght of stay, among others will be investigated.

DETAILED DESCRIPTION:
A prospective randomized clinical trial of all the patients undergoing Roux - en-Y gastric bypass will be performed. Patients will be randomly assigned into 2 groups: those patients receiving a preoperative balanced energy high-protein formula (group 1) and those receiving preoperative Immunonutrition (group 2). Changes between groups in acute inflamatory markers (CRP, fibrinogen, leucocites), pain (VAS scale), postoperative septic complications .(anastomotic leak and organ/space SSI)and lenght of stay, among others will be investigated.

ELIGIBILITY:
Inclusion Criteria:

1. Patients undergoing a laparoscopic gastric bypass (BPG) as a bariatric procedure
2. Men and Women older than 18 years.
3. Willing to participate in the study and giving their written consent

Exclusion Criteria:

1. Patients younger than 18 years.
2. Patients undergoing other bariatric surgery techniques.
3. Patients undergoing any other surgical procedure added to the bariatric technique.
4. Patients with medical or surgical pathologies that at the discretion of the investigator do not allow their participation in the study.
5. Inability to understand the nature and purpose of the study and / or to accept written participation in the study.
6. Impossibility to comply with pre-established clinical follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2016-02 (Actual); Primary Completion 2016-09 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Decrease in systemic inflamatory response in terms of CRP | 24h after surgery
  Proportion of patients with at least a 50% decrease in CRP 24 after surgery

SECONDARY OUTCOMES:
Decrease in systemic inflamatory response in terms of other inflamatory biomarkers | 24 hours after surgery
  Mean decrease in leukocite count, fibrinogen
Postoperative pain | 24h after surgery
  Mean VAS score
Complications | 30 days after surgery
  Rate of complications
In-hospital stay | 30 days after surgery
  In-hospital stay
Number of readmissions | 30 days after surgery
  Number of readmissions
Adverse Events Ocurrence | 30 days after surgery
  AE rate

CONTACTS AND LOCATIONS:
Overall Officials: Jaime Ruiz-Tovar, Principal Investigator — Fundacion Jimenez Diaz
Locations (1):
- Fundacion Jimenez Diaz, Madrid, Spain

REFERENCES:
- [Derived] Ruiz-Tovar J, Blanca M, Garcia A, Gonzalez J, Gutierrez S, Paniagua A, Prieto MJ, Ramallo L, Llanos L, Duran M. Preoperative administration of Omega-3 fatty acids on postoperative pain and acute-phase reactants in patients undergoing Roux-en-Y gastric bypass: A randomized clinical trial. Clin Nutr. 2019 Aug;38(4):1588-1593. doi: 10.1016/j.clnu.2018.07.026. Epub 2018 Jul 29. PMID 30097364